CLINICAL TRIAL: NCT04224415
Title: Re-challenge of Anti-EGFR Agents for Chinese Patients With RAS/BRAF Wild-type Metastatic Colorectal Cancer
Brief Title: Re-challenge of Anti-EGFR for Patients With RAS/BRAF Wild-type Metastatic CRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anti-EGFR Re-challenge
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C225+CPT-11 (Other): Patients will receive Systemic C225+CPT-11 every 14 days:
  C225 500 mg/m2 IV over 90 minutes on Day 1; Irinotecan 180 mg/m2 IV on Day 1
  Interventions: Drug: C225+CPT-11

INTERVENTIONS:
Drug: C225+CPT-11 — Patients will receive Systemic C225+CPT-11 every 14 days:
  C225 500 mg/m2 IV over 90 minutes on Day 1; Irinotecan 180 mg/m2 IV on Day 1

SUMMARY:
The aim of the trial is to study the efficacy and safety of Cetuximab re-challenge for Chinese Patients with RAS/BRAF wild-type Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
After first-line treatment of FOLFOX/FOLFIRI/FOLFOXIRI plus Cetuximab failure and defined as RAS/BRAF wild-type by molecular detection of cycle tumor DNA, the patients will be treated with Cetuximab and Irinotecan as a second-line or third-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤75.
* Diagnosed as colorectal adenocarcinoma by histology.
* Initially confirmed as RAS/BRAF wild type by tissue molecular detection.
* Treated with first-line therapy of FOLFOX/FOLFIRI/FOLFOXIRI+Cetuximab effectively and the PFS is not less than 6 months.
* Tumor progression during Cetuximab treatment or after treatment within 3 months.
* Tumor progression again after second-line treatment.
* The interval time of re-challenge is more than 4 months after the last time treated with Cetuximab.
* Lesions can be measured by the standard of RECIST v1.1.
* Defined as RAS/BRAF wild-type by molecular detection of cycle tumor DNA,
* No hematologic dysfunction(Platelets >90×10^9/L; WBC >3×10^9/L; Neutrophil >1.5×10^9/L；Hemoglobin >10 g/100ml).
* Serum bilirubin ≤ 1.5 × ULN; aminotransferase ≤ 5 × ULN.
* No ascites; no coagulation dysfunction; albumin ≥ 30g/L.
* Hepatic function was classified as class A by Child-Pugh classification.
* Serum creatinine < 1 × ULN, or creatinine clearance rate(CCR) > 50ml/ min(calculated by Cockcroft-Gault formula).
* ECOG scored as 0-2.
* Life expectancy > 3 months.
* Informed consent.
* Willing and able to receive follow-up until death or trial is finished or trial is terminated.

Exclusion Criteria:

* RAS/BRAF mutation.
* Severe arterial embolism or ascites.
* Presence of hemorrhagic tendency or coagulation dysfunction.
* Presence of hypertensive crisis or hypertensive encephalopathy.
* Severe uncontrolled systemic complications, such as infection or diabetes.
* Severe clinical CVD(cardiovascular disease), such as cerebrovascular accident(within 6 months before recruitment), myocardial infarction(within 6 months before recruitment), uncontrolled hypertension; unstable angina pectoris; congestive heart-failure(NYHA 2-4 grade); arrhythmia that needs medication treatment.
* Previous diagnosed or physical examination showed presence of central nervous system(CNS) disease(i.e. primary brain tumor, epilepsy uncontrolled by standard treatment, any history of brain metastases or stroke).
* Previous history of other malignancy within 5 years(except basal cell carcinoma after radical resection and/or cervical carcinoma in situ).
* Received any medication under research within 28 days before the trial.
* Any residual toxicity of previous chemotherapy(except hair loss), i.e. peripheral neuropathy ≥ NCI CTC v3.0 Grade 2, will be excluded from oxaliplatin-based chemotherapy regimen research pair.
* Allergic to any medication involved in the trial.
* Pregnant and lactating women.
* Patient who does not use or refuses to take any appropriate contraceptive measures (intrauterine contraceptive ring, barrier contraception combined with spermicidal gel or sterilization operation), including women of childbearing age (within 2 years after the last menstrual period) and men who are with possible fertility.
* Unable or unwilling to comply with the research plan.
* The existence of any other disease, dysfunction caused by metastatic lesions, or suspicious disease found on the regular examination, which indicating contraindications to the use of study drugs or may bring high risks of treatment related complications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 2-4 months
  defined as complete remission rates and partial remission rates after treatment.

SECONDARY OUTCOMES:
Progress-free Survival(PFS) | Up to 2-4 months
  defined as the period from the date of receiving treatment to disease progress caused by any reason.
Overall Survival(OS) | Up to 12 months
  defined as the period from the date of receiving treatment to death caused by any reason.
Adverse events(AE) and severe adverse events(SAE) | Up to 6 months
  defined as the incidence and severity of adverse events related to chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China